CLINICAL TRIAL: NCT04058119
Title: VIVE Mind: Terapias Corpo-mente Nos Cuidados de saúde primários - Estudo Aleatorizado e Controlado
Brief Title: Mind-Body Therapies in Primary Health Care
Acronym: VIVEmind
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidade de Saude da Ilha de Sao Miguel (Other)
Responsible Party: Principal Investigator, Sara B. Ponte, MD, General Practitioner, Unidade de Saude da Ilha de Sao Miguel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USISM_02_19
Record Dates: First submitted 2019-08-08; First posted 2019-08-15 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Psychological Stress
Keywords: Mind-body therapies; Yoga; Qigong; Pilates; Primary health care
MeSH Terms: conditions — Stress, Psychological | interventions — Mind-Body Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-body therapies (Experimental): Sessions of body-mind therapies (yoga, qigong and pilates)
  Interventions: Behavioral: Mind-body therapies
- Waiting list control group (No Intervention): Participants will not participate in any specific intervention, but will receive the Functional Training Program after the experimental period (6 months).

INTERVENTIONS:
Behavioral: Mind-body therapies — Sessions of body-mind therapies (yoga, qigong and pilates), oriented by certified instructors. Every sessions will be 60-minutes long, biweekly, with a total duration of 6 months.
  Arms: Mind-body therapies

SUMMARY:
Mental disorders are among the most common causes of disability globally. Given the high prevalence of mental disorders (57.0%) in Azores islands (Portugal), local primary health care (PHC) services should encourage the implementation of complementary interventions for prevention of this type of disorders. New approaches, such as mind-body therapies, have been studied and recommended for prevention and treatment of numerous chronic diseases, particularly mental disorders.

This study aims to evaluate the feasibility and effectiveness of a 6-months mind-body therapies (yoga, qigong and pilates), in users of Ponta Delgada Health Center (PDHC) with perceived distress, compared to a waiting list control.

DETAILED DESCRIPTION:
VIVE mind will be a pragmatic, single-center, randomized controlled trial.

Users of PDHC with perceived distress (PSS-10), aged 18 years or over, will be recruited and randomly assigned into experimental and waiting list control group, in a 1:1 ratio. The recruitment of participants will be held in PDHC by health professional (e.g., family medicine doctors, nurses, nutritionists, psychologists, etc). After signed informed consent and baseline measures, experimental group will participate in body-mind sessions (yoga, qigong or pilates), oriented by certified instructors, during 6-months. Each participant should attend only one of the therapies, in order to guarantee a differentiated evaluation. In every session, it will be evaluated the participants' adherence and theirs perceived enjoyment and exertion. The other outcomes (primary and secondary) will be analyzed through a face-to-face contact, in three different moments: baseline (T0), post-intervention (at month 6, T1) and 6-month follow-up (at month 12, T2). The control group will not participate in any specific intervention, but will receive the body-mind intervention after the experimental period. An intention-to-treat and per protocol analysis will be performed to analyze intervention effectiveness and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Users of Ponta Delgada Health Center with perceived distress (score higher than 20 for men and higher than 22 for women in PSS-10).

Exclusion Criteria:

* Users with recent practice (less than 3 months) of any mind-body therapies;
* Users with medical contraindications to moderate-to-vigorous intensity physical activities, such as: unstable angina; deep vein thrombosis; recent thromboembolism or embolism; acute systemic infection or fever; atrioventricular block of 2nd grade or higher (without pacemaker); negative deflection of the ST segment deflection of the ST segment > 2 mm; severe neuro-musculoskeletal dysfunction; severe mitral or aortic insufficiency or stenosis without adequate treatment; decompensated heart failure; resting heart rate above 100 bpm; other decompensated metabolic disorders; pericarditis or acute myocarditis; uncontrolled arrhythmia; uncontrolled resting hypertension (SBP ≥ 180 or DBP ≥ 110); orthostatic hypotension with a fall in SBP> 20 mmHg or uncontrolled diabetes;
* Users with physical and/or mental disabilities;
* Users with severe psychiatric diagnosis or/and active psychosis or
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Perceived Stress Scale (PSS 10), validated for portuguese population, is a self-report scale with 10 items on daily hassles and the current feeling of being able to handle problems that need to be addressed. It is a five-point Likert scale ranging from 0 (never) to 4 (very often). This questionnaire is widely used to measure perceived stress and has adequate internal and test-retest reliability.

SECONDARY OUTCOMES:
Adherence to the mind-body sessions | Up to 6 months
  Proportion of adherence to the mind-body sessions will be calculated by the average of adherence of each participant. The adherence of each participant will be quantified by the relationship between the sessions attended and the total number of sessions scheduled over the 6 months.
Perceived enjoyment | Up to 6 months
  Perceived enjoyment of the mind-body sessions will be measured biweekly by a scale rated from 1 (very unpleasant) to 5 (very enjoyable).
Perceived exertion | Up to 6 months
  Perception exertion of mind-body sessions will be measured biweekly by the modified Borg scale. In this instrument, 11 items are evaluated, with a score of 0 to 10 points, where 0 equals the minimum effort and 10 the maximum that they can perform.
Participants' satisfaction | T1, Post-intervention (at month 6)
  Participant's satisfaction levels will be measured by 10-items questionnaire, on a five point Likert scale from 1 (displeased) to 5 (very satisfied).
Change in hand grip strength | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Hand grip strength will be evaluated while the participant is in a sitting position with shoulders adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral and wrist between 0 and 30° of extension. The test will be repeated 3 times with the dominant hand, and maximum reading will be taken.
Change in body mass index (BMI) | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Weight (kilograms) and height (meters) will be combined to report BMI in kg/m^2.
Change in waist circumference | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Waist circumference in centimeters.
Change in body fat | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Measured by bioelectrical impedance analysis.
Change in body lean mass | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Measured by bioelectrical impedance analysis.
Change in systolic and diastolic blood pressure | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Resting systolic blood pressure.
Change in fast blood glycemia | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Fast blood glycemia (mg/dL).
Change in HbA1c | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  HbA1c (%) reflects the average plasma glucose over the previous 8 to 12 weeks.
Change in blood lipid profile | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides.
Change in chronic pain | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Brief Pain Inventory (BPI) will assess the average pain at rest, using a numerical (0-10) rating scale on the BPI Short Form. A higher score indicates worse pain (10 is "worst pain imaginable") and zero indicates 'no pain at all'.
Change in nicotine dependence | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Fagerström Test for Nicotine Dependence (FTND) will be applied only in smokers participants.
  FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Change in analgesic and psychotropic medication dependence | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Number of analgesic and psychotropic pills ingested per day.
Change in health-related quality of life | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  The health-related quality of life questionaire EQ-5D-5L is a standardised self-report measure of health status developed by the EuroQol Group. It consists of the descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions, namely mobility, self care, usual activities, pain/discomfort, anxiety/depression.
Change in psychological distress | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Depression, anxiety stress scale-21 (DASS-21) consists of three 7-item subscales: depression, anxiety, and stress. Participants indicate how much each of 21 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). This scale has good psychometric properties in both clinical and non-clinical samples. Also, this scale reliably distinguishes between symptoms of anxiety (panic/worry), stress (tension/agitation) and depression (low mood/anhedonia), which are highly comorbid.
Change in mental well-being | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item scale, validated and self-report instrument used to assess mental wellbeing in general population. Possible scores range from range from 14-70, with higher scores indicating higher mental well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Sara B. Ponte, MD, Principal Investigator — Unidade de Saúde da Ilha de São Miguel
Locations (1):
- Centro de Saúde de Ponta Delgada (Unidade de Saúde da Ilha de São Miguel), Ponta Delgada, Azores, Portugal